CLINICAL TRIAL: NCT06481618
Title: Impact of Stress the Management of BAVU Ventilation (Self-filling Bag With One-way Valve) by Healthcare Professionals.
Brief Title: Impact of Stress on Management of BAVU Ventilation (Self-filling Bag With One-way Valve) by Healthcare Professionals.
Acronym: SIMBAVU 2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2024 GODET (SIMBAVU 2); 2024-A00919-38 (Other: 2024-A00919-38)
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-06

CONDITIONS: Any Healthcare Professional; Agreement to Participate; Who May be Required to Perform Manual Ventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the impact of stress on the manual ventilation through Self-filling Bag With One-way Valve. The main question it aims to answer :

how does the ocurence of a stressfull event modify the ventilation delivered in term of pressure, frequency, volume.

Volunter healthcare professionals will take part in a simulation where they will manually ventilate a manikin and ventilation datas will be recorded.

DETAILED DESCRIPTION:
The lung simulator (ASL 5000TM, IngMar Medical) will be connected to a high-fidelity mannequin (SimMan 3G, Laerdal Medical). A continuous, cycle-by-cycle recording of the administered ventilatory parameters will be carried out (recording of pressure, volume and flow curves as a function of time). These curves will then make it possible to determine the main parameters of this ventilation (respiratory frequency, maximum and end-expiratory pressure, tidal volume, etc.).

The healthcare professional will be asked to carry out ventilation with Self-filling Bag With One-way Valve as he is accustomed to doing, during a standardized patient transfer.

Subsequently, an unforeseen event will be added to the situation with continued continuous recording of ventilation modalities.

The personal data that will be requested from healthcare professionals will be: their age, their gender, their seniority in the profession, their place of practice. The stress of healthcare professionals will be assessed using a digital self-assessment scale and the use of a heart rate monitor.

Prior stress and anxiety will be measured in advance by completing several questionnaires before starting the simulation (STAI-T, STAI E, AD ACL).

ELIGIBILITY:
Inclusion Criteria:

* Any healthcare professional who may be required to perform manual ventilation

Exclusion Criteria:

* Unavailability of simulation equipment
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any healthcare professional who may be required to perform manual ventilation with Self-filling Bag With One-way Valve, available to participate in this work and not opposed to their inclusion in this study.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
ventilation quality | 1 hour
  Quality of ventilation under stress conditions in terms of frequency, pressure and volume delivered compared to the standards of the protective ventilation initially delivered

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Godet, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France